CLINICAL TRIAL: NCT05697315
Title: The Effect of Erector Spinae Block for Postoperative Pain Management Cesarean Delivery Patients
Brief Title: Erector Spinae Plane Block for Postoperative Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Gökçe Gişi, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-02-03
Record Dates: First submitted 2023-01-04; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Pain; Post Operative Pain
Keywords: Pain; postoperative analgesia; Erector spinae plane block; cesarean section
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double (Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): No block was performed, tramadol was administered with patient-controlled analgesia (PCA) and all patients were followed in the ward.
  Interventions: Procedure: Control
- Erector spinae plane block (Active Comparator): Erector spinae plane block was performed, tramadol was administered with patient-controlled analgesia (PCA) and all patients were followed in the ward.
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Control — No block was performed
  Arms: Control group
Procedure: Erector spinae plane block — Erector spinae plane block was performed, tramadol was administered with patient-controlled analgesia (PCA) and all patients were followed in the ward.
  Arms: Erector spinae plane block

SUMMARY:
Erector spinae plane (ESP) block is an interfacial plane block with visceral and somatic analgesic activity at paraspinal muscles. This study aims to examine the postoperative analgesic efficacy of ESP block after cesarean section (CS) with Pfannenstiel incision under spinal anesthesia.

DETAILED DESCRIPTION:
The study included 54 patients with mild systemic disease (ASA II patients) who would undergo elective CS under spinal anesthesia. They were randomly divided into an ESP block group (Group E) and a control group (Group C). After the surgery, Group E patients underwent ultrasound-guided bilateral ESP block with 20 ml of 0.25% bupivacaine at the lateral decubitus position, while Group C received no intervention. Patients in both groups received parenteral patient-controlled analgesia. The patients' post-operative 24-hour opioid consumption, regular Visual Analogue Scale (VAS) measurements, and need for rescue analgesics were evaluated. Statistical analysis was performed using SPSS 21 program. Demographic and other data were assessed using independent samples t-test, Mann-Whitney U test, and Chi-square analysis.

ELIGIBILITY:
Inclusion Criteria:

* ASA II patients
* 18-45 years who underwent CS with Pfannenstiel incision under spinal anesthesia
* agreed to participate in the study

Exclusion Criteria:

* Patients with infection at the injection site
* Coagulopathy Allergy to amide-type local anesthetics
* History of peripheral neuropathy
* Hepatic and/or renal failure
* Refusing the procedure
* patients with heart disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 56 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
24-hour opioid consumption | up to 24 hour
  The amount of tramadol consumed in milligrams in the first 24 hours was determined with a patient-controlled analgesia pump.

SECONDARY OUTCOMES:
Visual Analog Scale (Vas) | 0, 30 minutes, 1 hour, 2 hours, 6 hours, 12 hours, 24 hours
  pain scores,graded from 0 to 10, 0 no pain, 10 highest pain experienced

CONTACTS AND LOCATIONS:
Overall Officials: Gökçe Gişi, Principal Investigator — Kahramanmaras Sutcu Imam University Hospital Kahramanmaras, Turkey
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided